CLINICAL TRIAL: NCT05293106
Title: Assessing the Hemostatic Efficacy of Pathogen Reduced Platelets in Children Undergoing Cardiopulmonary Bypass Surgery: A Pilot Clinical Trial
Acronym: PEDITREC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting and enrolling subjects.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-11024115
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Cardiopulmonary Bypass Surgery
Keywords: Platelet Transfusion; LVDS platelet transfusion; PR platelet transfusion
MeSH Terms: interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pathogen-reduced (PR) platelet transfusions (Active Comparator): FDA approved and already used in this patient population
  Interventions: Biological: Platelet Transfusion
- Large volume delayed sampling - LVDS (Active Comparator): FDA approved and already used in this patient population
  Interventions: Biological: Platelet Transfusion
- No platelet transfusion (No Intervention): Subject will not receive a platelet transfusion

INTERVENTIONS:
Biological: Platelet Transfusion — All platelet transfusions will be given as 10mL/kg as is considered standard of care.
  Arms: Large volume delayed sampling - LVDS; Pathogen-reduced (PR) platelet transfusions

SUMMARY:
This study is testing whether pathogen reduced platelets can control bleeding as well as non-pathogen reduced platelets (otherwise known as large volume delayed sampling).

DETAILED DESCRIPTION:
This is a pilot clinical trial to assess the post-operative bleeding in children who receive pathogen-reduced (PR) platelet transfusions versus standard (large volume delayed sampling - LVDS) platelet transfusions both during and for 24 hours following cardiopulmonary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 0 up to and including 18 years of age
* Undergoing elective cardiopulmonary bypass surgery
* Are planned to have a chest tube placed in the operating room prior to chest closure

Exclusion Criteria:

* >/=19 years of age
* Preterm infants (less than 38-week gestational age at time of surgery)
* On extracorporeal membrane oxygenation (ECMO) or ventricular assist device prior to surgery
* Family requests limitation of blood products (i.e. Jehovah's Witness)
* Congenital bleeding disorder
* Are planned to require ECMO post-op
* Previously enrolled in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Nellis, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Morgan Stanley Children's Hospital at Columbia University, New York, New York
  - Komansky Children's Hospital at Weill Cornell, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric patients were recruited in the pre-operative cardiology clinic from 6/1/2022-12/31/2023 at Komansky Children's Hospital at Weill Cornell.
  For neonates admitted for their birth and awaiting cardiac surgery, the families were approached approached in the neonatal intensive care unit by the CT surgery team.
Period: Overall Study
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Started | 1 | 1 | 7
Completed | 1 | 1 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion | Total
Number analyzed (Participants) | 1 | 1 | 7 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: months] — in months (of note if patient's age is less than one month, it is noted as 0)
  months | 0 [0 to 0] | 72 [72 to 72] | 117 [48 to 181] | 81 [48 to 132]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 5 | 5
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 2
  Black | 0 | 0 | 1 | 1
  White | 1 | 0 | 4 | 5
  Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Bleeding Measured by Chest Tube Output for First 24 Hours Following Cardiopulmonary Bypass Surgery
Description: Chest tube output for first 24 hours following cardiopulmonary bypass surgery
Time Frame: Within the first 24 hours post-op.
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Number analyzed (Participants) | 1 | 1 | 7
mL/kg | 35.3 [35.3 to 35.3] | 21.0 [21.0 to 21.0] | 6.6 [5.1 to 10.5]

2. Secondary Outcome: Total Dose Red Blood Cell Volume Transfused in First 48 Hours Post-op
Description: Total dose red blood cell volume transfused in first 48 hours post-op (includes both red blood cell as well as cellsaver)
Time Frame: During hospitalization in the first 48 hours (no follow-up visits necessary)
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Number analyzed (Participants) | 1 | 1 | 7
mL/kg | 18.8 [18.8 to 18.8] | 20.3 [20.3 to 20.3] | 4.8 [0 to 6.3]

3. Secondary Outcome: Total Platelet Volume Transfused in the First 48 Hours Post-op
Description: Total platelet volume transfused in the first 48 hours post-op
Time Frame: During hospitalization in the first 48 hours (no follow-up visits necessary)
Population: This Outcome Measure was not assessed in the No Platelet Transfusion Arm/Group
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Number analyzed (Participants) | 1 | 1 | 0
mL/kg | 18.8 [18.8 to 18.8] | 14.1 [14.1 to 14.1] |

4. Secondary Outcome: Total Plasma Volume Transfused in the First 48 Hours Post-op
Description: Total plasma volume transfused in the first 48 hours post-op
Time Frame: During hospitalization in the first 48 hours (no follow-up visits necessary)
Population: This Outcome Measure was not assessed in the No Platelet Transfusion Arm/Group
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Number analyzed (Participants) | 1 | 1 | 0
mL/kg | 18.1 [18.1 to 18.1] | 10 [10 to 10] |

5. Secondary Outcome: Total Cryoprecipitate Volume Transfused in the First 48 Hours Post-op.
Description: Total cryoprecipitate volume transfused in the first 48 hours post-op.
Time Frame: During hospitalization in the first 48 hours (no follow-up visits necessary)
Population: This Outcome Measure was not assessed in the No Platelet Transfusion Arm/Group
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
Number analyzed (Participants) | 1 | 1 | 0
mL/kg | 17.5 [17.5 to 17.5] | 5.1 [5.1 to 5.1] |

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the subjects hospital course (varied by patient but no longer than 14 days)
Arm/Group | Pathogen-reduced (PR) Platelet Transfusions | Large Volume Delayed Sampling - LVDS | No Platelet Transfusion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/7

LIMITATIONS AND CAVEATS:
Due to difficulty in recruiting and enrolling subjects, only descriptive statistics were used to describe the 9 enrolled subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT05293106/Prot_SAP_000.pdf